CLINICAL TRIAL: NCT04969770
Title: Contribution of Muscle and Disc Elastography in the Evaluation of Biomechanical Modifications of the Neuromuscular Spine Fixed by Bipolar Construct
Brief Title: Evaluation of Biomechanical Modifications of the Neuromuscular Spine Fixed by Bipolar Construct
Acronym: ELASTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210752; ID-RCB 2020-A03598-31 (Other: ID-RCB Number)
Record Dates: First submitted 2021-06-25; First posted 2021-07-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Neuromuscular Scoliosis
Keywords: Neuromuscular scoliosis; Innovative fusionless surgery; Bipolar spine construct; Minimally invasive approach; Ultrasound elastography (USE)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neuromuscular scoliosis (Experimental): Minor patients with neuromuscular scoliosis and followed at Necker Hospital
  Interventions: Other: Ultrasound elastography (USE)
- Neuromuscular pathologies without instrumented scoliosis (Other): Minor patients with neuromuscular pathology without instrumented scoliosis and followed at Necker Hospital
  Interventions: Other: Ultrasound elastography (USE)
- Controls (Other): Minor patients without neuromuscular pathology or scoliosis and followed at Necker Hospital
  Interventions: Other: Ultrasound elastography (USE)

INTERVENTIONS:
Other: Ultrasound elastography (USE) — Visualization of the vertebral disc and the para-vertebral muscles.
  Intra and inter observer reproducibility analysis carried out for each of the measurements made, by two operators.
  Patients with instrumented neuromuscular scoliosis: 5 elastographies : preoperatively, then during the usual follow-up consultations with the surgeon every 6 months for 2 years.
  Patients with neuromuscular pathologies without instrumented scoliosis: 4 elastographies during the usual follow-up consultations with the surgeon every 6 months for 2 years.
  Healthy control patients without neuromuscular pathology or scoliosis :
  1 elastography during an usual consultation.

SUMMARY:
Neuromuscular scoliosis are caused by a disorder of the brain, spinal cord or muscular system and often progressive at early age. Conservative treatment is not sufficient to maintain trunk and pelvic balance, and surgical treatment is frequently required. Early definitive spine fusion has the disadvantage of cessation of trunk growth with concomitant effects on lung development. Growth preserving spine surgeries are increasingly used but with high complication rates.

The orthopaedic team at Necker Hospital Enfants maladies, Paris, France has developed an innovative fusionless surgery based on a bipolar spine construct, performed by a minimally invasive approach. The first 100 patients operated on with this technique had an average follow-up of 6.5 years. No arthrodesis, initially planned in adolescence, was necessary thanks to the stability of the correction of the deformities even after skeletal maturation.

The main objective of the study was to analyze the progressive spinal stiffening, using muscle and disc elastography, in neuromuscular patients instrumented with this bipolar construct.

DETAILED DESCRIPTION:
Neuromuscular scoliosis is related to muscle tone abnormalities with a prognosis worsen by damage to the axial and respiratory muscles.

The classic treatment for these scoliosis consists of conservative treatment (physiotherapy, bracing), followed by arthrodesis in adolescence. Arthrodesis consists of a global posterior spinal fusion, with a high risk of septic and hemorrhagic complications.

In cases of early and rapidly progressive deformities, fusionless techniques allow the preservation of growth while waiting for arthrodesis. However, these techniques have a high rate of complications, particularly of mechanical and infectious origin, which led the orthopedic team at Necker Hospital, Paris, France to develop an innovative technique. This technique is based on bipolar construct, performed by a minimally invasive approach. The first 100 patients operated on have an average follow-up of 6.5 years. No arthrodesis, initially planned in adolescence for these patients, was necessary, thanks to the stability of the correction even after skeletal maturation.

The main objective of the study was to analyze the progressive spinal stiffening, using muscle and disc elastography, in neuromuscular patients instrumented with this bipolar construct.

ELIGIBILITY:
Inclusion Criteria:

* Minor patients between 10 and <18 years old, presenting a neuromuscular pathology, with progressive scoliosis, to undergo for their clinical care a fusionless surgery based on a bipolar spine construct, performed by a minimally invasive approach
* Minor patients between 10 and <18 years old, presenting a neuromuscular pathology such as encephalopathy / infantile spinal amyotrophy / myopathy, without progressive scoliosis
* Minor patients between 10 and <18 years old, healthy controls, followed in orthopedics for a pathology other than neuromuscular or spinal deformity
* Written informed consent

Exclusion Criteria:

* No social insurance
* Severe mental retardation or severe dystonia making data acquisition impossible or requiring sedation
* Patients with gastrostomy or tracheostomy

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Discal stiffness | 2 years
  Ultrasound elastography (USE) Measurements performed in the transverse plane of L3-L4 intervertebral disc. A rectangular strip is selected and a series of 3 clips of 10 seconds (i.e., 30 images) is recorded. The average of these measurements is reported.
Paravertebral muscular stiffness | 2 years
  Ultrasound elastography (USE) Measurement performed in the longitudinal plane, in the axis of muscular fibers and in the middle of multifidus muscle.
  A rectangular strip is selected and a series of 3 clips of 10 seconds (i.e. 30 images) is recorded. The average of these measurements is reported in rest and passive stretching position, on the right side and on the left side.

SECONDARY OUTCOMES:
Parameters influencing the progressive stiffening of the spine | 2 years
  Research and description of clinical parameters influencing the progressive stiffening of the spine, e.g. , age, etiology, spinal deformity and correction, BMI
Biomechanical characteristics of the construct | 2 years
  Influence of spinal stiffness on biomechanical characteristics of the construct : distance between the rods and the spine, causing an osteo-inductive process
Occurrence of rod fracture | 2 years
  Occurrence or not of a rod fracture on X-rays

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Gaume, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Lofti Miladi, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaume M, Loiselet K, Chekir H, Langlais T, Boddaert N, Stricker S, Pannier S, Skalli W, Miladi L, Vergari C. Evidence of spinal stiffening following fusionless bipolar fixation for neuromuscular scoliosis: a shear wave elastography assessment of lumbar annulus fibrosus. Eur Spine J. 2024 Apr;33(4):1617-1623. doi: 10.1007/s00586-023-08013-8. Epub 2023 Nov 4. PMID 37924389